CLINICAL TRIAL: NCT05783947
Title: Diagnostic Performance of a Commercial Indirect Immunofluorescence Assay for the Detection of Neuronal Antibodies in Auto-immune Encephalitis and Paraneoplastic Neurological Syndromes
Brief Title: Diagnostic Performance of a Commercial Assay for the Detection of Neuronal Antibodies
Acronym: IFINEURO
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 23-5024
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Paraneoplastic Neurological Syndrome; Autoimmune Encephalitis
Keywords: autoantibodies; diagnostic; paraneoplastic; encephalitis; neuronal
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System; Disease; Encephalitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum and CSF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspicion of autoimmune neurological disorder: Sera and CSF of patients with a suspicion of autoimmune encephalitis or paraneoplastic neurological syndrome
  Interventions: Diagnostic Test: Indirect immunofluorescence assay on tissue slides and cell-based assays with CSF and/or sera

INTERVENTIONS:
Diagnostic Test: Indirect immunofluorescence assay on tissue slides and cell-based assays with CSF and/or sera — Sera and/or CSF samples are drawn from patients with a clinical suspicion of autoimmune encephalitis or paraneoplastic neurological syndrome. Indirect immunofluorescence assays will be performed on commercial and in-house slides upon receipt in our center. In case of positive staining, additional tests such as cell-based assays, western-blots, ELISA or immunodots can be performed.

SUMMARY:
Detection of autoantibodies targeting neuronal surface or intracellular antigens is a keystone for the diagnosis and the treatment of auto-immune encephalitis and paraneoplastic neurological syndromes. A strategy commonly used for their detection is to perform a screening with a tissue-based immunofluorescence assay or immunohistochemistry assay and a second line test to confirm and identify the autoantibody. Since several years, commercial kits are used by a growing number of laboratories to screen the presence of these autoantibodies. However, the diagnostic performance of these commercial kits is highly variable and several studies reported a high prevalence of false-positive and false-negative results with commercial immunodots and cell-based assays. It is therefore essential to explore commercial kits limitations in order to avoid false-positive and false-negative results that could lead to misdiagnosis and/or to delay the treatments.

To assess the diagnostic performance of commercial kits, the investigators performed a prospective study in which the investigators screened patients neuronal autoantibodies in cerebrospinal fluid and sera using commercial tissue-based indirect immunofluorescence assay and CBAs in comparison with an in-house tissue-based indirect immunofluorescence assay.

ELIGIBILITY:
* Inclusion Criteria * : Sera and/or CSF with sufficient volume to perform both in-house and commercial assays
* Exclusion Criteria * : Sera and/or CSF with insufficient volume to perform both in-house and commercial assays

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a suspicion of autoimmune encephalitis or paraneoplastic neurological syndrome
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Number of discrepant results between commercial and in-house assays | at the baseline
  Both in-house and commercial assays will be performed independently and results will be compared once all tests are done. Number of discrepant results will be compared with concordant results according to the autoantibody identified.

CONTACTS AND LOCATIONS:
Overall Officials: Jérome HONNORAT, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - Hospice Civils de Lyon, Bron
  - Hospices Civils de Lyon, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: No